CLINICAL TRIAL: NCT00022347
Title: A Phase II Study of TLK 286 in Platinum Resistant Advanced Epithelial Ovarian Cancer
Brief Title: TLK286 in Treating Patients With Advanced Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: TLK-286.2003; MSKCC-01059; CDR0000068807 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1998
Record Dates: First submitted 2001-08-10; First posted 2004-01-14 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — TER 286

INTERVENTIONS:
Drug: canfosfamide hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of TLK286 in treating patients who have advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate and disease stabilization rate in patients with platinum-resistant advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer treated with TLK286. II. Determine the safety of this regimen in these patients. III. Determine the duration of objective response, time to tumor progression, and overall survival in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive TLK286 IV over 30 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks for 1 year and then every 12 weeks thereafter.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed advanced ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cancer Serous papillary Endometrioid Mucinous Clear cell Poorly differentiated adenocarcinomas Mixture of any of the above histologies No sarcomatous, stromal, or germ cell elements Measurable disease by radiological imaging with progression in the past 3 months or no response to prior therapy The following are not considered measurable: Pleural effusions Ascites Osseous metastases CA-125 tumor markers Lesions in previously irradiated areas Platinum resistant or refractory Less than 6 month treatment-free interval after platinum-containing regimen OR Progression during platinum-based therapy No leptomeningeal or carcinomatous meningitis Known CNS metastases allowed if patient is previously treated, neurologically stable, has no evidence of active disease by CT or MRI, and has no requirement for therapy with oral or IV steroids or anticonvulsants

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9.0 g/dL Hepatic: Bilirubin no greater than 2.5 mg/dL ALT and AST no greater than 3.0 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min No gross hematuria Cardiovascular: No uncontrolled cardiac arrhythmia No myocardial infarction within the past 6 months Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 6 months after study No unstable medical conditions No severe concurrent disease or infection that would preclude study No intestinal obstruction interfering with nutrition No psychiatric disorders that would preclude study No other prior malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy and recovered At least 2 weeks since prior prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF) No concurrent immunotherapy No concurrent biological response modifiers Chemotherapy: See Disease Characteristics At least 1 but no more than 3 prior chemotherapy regimens (platinum-containing regimens count as 1 regimen) At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: At least 4 weeks since prior radiotherapy or radiopharmaceuticals and recovered No prior radiotherapy to whole pelvis No concurrent radiotherapy including palliative radiotherapy (except local radiotherapy for pain or solitary brain metastasis if not progressing systemically) Surgery: At least 4 weeks since prior major surgery and recovered Other: At least 30 days since prior investigational drugs No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2004-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate
Safety
Duration of objective response
Time to tumor progression
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spriggs, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Kavanagh JJ, Gershenson DM, Choi H, Lewis L, Patel K, Brown GL, Garcia A, Spriggs DR. Multi-institutional phase 2 study of TLK286 (TELCYTA, a glutathione S-transferase P1-1 activated glutathione analog prodrug) in patients with platinum and paclitaxel refractory or resistant ovarian cancer. Int J Gynecol Cancer. 2005 Jul-Aug;15(4):593-600. doi: 10.1111/j.1525-1438.2005.00114.x. PMID 16014111